CLINICAL TRIAL: NCT03848130
Title: Effects of Lateral Wedge Insoles, Knee Taping on the Management of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Rabbiya Riaz, Physiotherapist, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIRS-1509/PDPT/010
Record Dates: First submitted 2019-01-25; First posted 2019-02-20 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Medial Compartment Knee Osteoarthritis
Keywords: Knee osteoarthritis; Knee injury and Osteoarthritis Outcome Score; Rapid assessment of physical activity; Quality of life; Traditional physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Knee Taping with Home Exercises (Group 1) (Active Comparator): Knee osteoarthritis patients were assessed by general demographic questionnaire, rapid assessment of physical activity (RAPA) to determine physical activity level and Knee injury and Osteoarthritis Outcome Score (KOOS) to determine the level of pain severity,stiffness, functional activities, recreational activities and Quality of life for enhancing functional independence and were assigned into knee taping group.Each subject in first group completed 4 weeks of physical therapy sessions which were aimed to decrease pain and stiffness, increase functional activity level, and improve quality of life. Each subject was evaluated for changes in symptoms on, 1st week, 2nd week, 3rd week and 4th week.
  Interventions: Other: Mulligan Knee Taping with Home Exercises
- Lateral wedge insoles with Home Exercises (Group 2) (Active Comparator): Knee osteoarthritis patients were assessed by general demographic questionnaire, rapid assessment of physical activity (RAPA) to determine physical activity level and Knee injury and Osteoarthritis Outcome Score (KOOS) to determine the level of pain severity,stiffness, functional activities, recreational activities and Quality of life for enhancing functional independence and were assigned into lateral wedge insole group.Each subject in second group completed 4 weeks of physical therapy sessions which were aimed to decrease pain and stiffness, increase functional activity level, and improve quality of life. Each subject was evaluated for changes in symptoms on, 1st week, 2nd week, 3rd week and 4th week.
  Interventions: Other: Lateral wedge insoles with Home Exercises
- Traditional Physiotherapy with Home Exercises (Group 3) (Active Comparator): Knee osteoarthritis patients were assessed by general demographic questionnaire, rapid assessment of physical activity (RAPA) to determine physical activity level and Knee injury and Osteoarthritis Outcome Score (KOOS) to determine the level of pain severity,stiffness, functional activities, recreational activities and Quality of life for enhancing functional independence and were assigned into traditional physiotherapy group.Each subject in third group completed 4 weeks of physical therapy sessions which were aimed to decrease pain and stiffness, increase functional activity level, and improve quality of life. Each subject was evaluated for changes in symptoms on, 1st week, 2nd week, 3rd week and 4th week.
  Interventions: Other: Traditional Physiotherapy with Home Exercises

INTERVENTIONS:
Other: Mulligan Knee Taping with Home Exercises — Each patient in group I i.e. taping group with home exercises was given 40 minutes session. Each session started in sitting or lying position with leg extended and mulligan tape was used. Taping was started in the middle of patella, at the level of superior aspect of patella and pulled the tape medially and fixed the tape at medial border. This tilts the lateral border of patella away from femur and produced skin wrinkling. Besides this, home exercises such as quads isometrics and self stretchings & ROMs were also guided. This session was repeated three times a week for one month (Total 12 sessions/ one month).
  Arms: Knee Taping with Home Exercises (Group 1)
Other: Lateral wedge insoles with Home Exercises — Each patient in group II i.e. lateral wedge insole with home exercises group was given 20-minute session. In each session, Lateral wedge insoles of 7mm made of silicon or ledos material were advised and home exercises in the same way. This session was repeated once a month but evaluations were obtained after a complete week for one month. (Total 4 sessions/one month)
  Arms: Lateral wedge insoles with Home Exercises (Group 2)
Other: Traditional Physiotherapy with Home Exercises — Each patient in group III i.e. traditional physiotherapy with home exercises group was given 40 to 45-minute session. Each session started in lying position. In each session, therapeutic ultrasound with 1.5MHz frequency and continuous mode for 7 minute was given. Then passive stretchings of the following muscle groups was done; calf, hamstring, quadriceps, hip flexors and hip adductors & abductors and followed by strengthening exercises manually and with quadriceps bench. Home exercises were guided in the same way. This session was repeated 3 to 4 times a month. (Total 12 to 16 sessions/ one month)
  Arms: Traditional Physiotherapy with Home Exercises (Group 3)

SUMMARY:
Knee osteoarthritis (OA) is a degenerative, progressive and wide spread disease, which may lead the patient to severe outcomes e.g. pain, loss of joint motion, inflexibility, disability and decreases the quality of life (QOL). As it affects the adults of older age, therefore should be emphasized.Effectiveness of Mulligan knee taping, lateral wedge insoles and traditional physical therapy(Ultrasound therapy with stretching and strengthening exercises) with home exercises as baseline treatment were assessed through RAPA and complete KOOS questionnaire.

DETAILED DESCRIPTION:
A total of 60 patients with medial compartment 3rd grade knee osteoarthritis were recruited and randomly divided into three groups, 20 in each group.The data was collected through general demographic questionnaire, rapid assessment of physical activity (RAPA) to determine physical activity level and Knee injury and Osteoarthritis Outcome Score (KOOS) to determine the level of pain severity, stiffness, functional activities, recreational activities and Quality of life for enhancing functional independence while having osteoarthritis. For between-group analysis, one way ANOVA was used and for within-group analysis longitudinal repeated measures analysis of variance (RM-ANOVA) with Tukey's multiple comparisons test was used.

ELIGIBILITY:
Inclusion Criteria:

* Knee OA in the age group of 40-70 year.
* Knee OA due to aging.
* Knee OA due to family history

Exclusion Criteria:

* Knee OA due to Trauma.
* Knee OA due to any knee pathology.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Knee injury and osteoarthritis outcome pain score | Upto 4 weeks
  Pain associated with daily tasks is measured through Knee injury and osteoarthritis outcome pain score scale with categories as "None" for no pain and "Extreme" for maximum pain value.
Knee injury and osteoarthritis outcome stiffness score | Upto 4 weeks
  It is also measured through Knee injury and osteoarthritis outcome stiffness score scale with categories as "None" for no pain and "Extreme" for maximum pain value.
Knee injury and osteoarthritis outcome functional status score | Upto 4 weeks
  Degree of difficulty in performing daily tasks associated with knee joint is measured through Knee injury and osteoarthritis outcome functional status score in categories as "None" for no difficulty in task and "Extreme" for maximum difficulty in performing task.
Knee injury and osteoarthritis outcome quality of life score | Upto 4 weeks
  Quality of life regarding knee joint disease is measured through Knee injury and osteoarthritis outcome quality of life score in categories as according to patient's satisfaction.

SECONDARY OUTCOMES:
Rapid Assessment Physical Activity scale | Upto 4 weeks
  Physical activity level of the patients was also observed through rapid assessment of physical activity with categories as "0" for No involvement and "1" for yes and the results showed that those who are involved in any type of physical activity have a better functional outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabbiya Riaz, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR